CLINICAL TRIAL: NCT02627703
Title: A Prospective Clinical Utility Study of the Impact of the 21 Gene Recurrence Score® Assay (Oncotype DX®) in Estrogen Receptor Positive (ER+) HER-2 Negative (HER 2-) 1-3 Node Positive (pN1) Breast Cancer in Multiple BC Cancer Agency Centres
Brief Title: (Oncotype DX®) in Estrogen Receptor Positive (ER+) HER-2 Negative (HER 2-) 1-3 Node Positive (pN1) Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: Genomic Health®, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 01-168
Record Dates: First submitted 2015-11-23; First posted 2015-12-11 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Oncotype DX — The Oncotype DX® assay is a multi-gene reverse-transcriptase-polymerase-chain-reaction (RT-PCR) test that analyzes the expression of 21 genes, and quantifies the 10 year distant breast cancer recurrence risk in patients with stage I and II, lymph node negative, estrogen receptor positive disease who plan to be treated with tamoxifen for 5 years.

SUMMARY:
This study is a multi-center BCCA study that evaluates the impact of the Oncotype DX® assay on the decision making of the treating physician and the patient. The Oncotype DX® assay is a commercially available diagnostic test that aids in a physician's treatment recommendation to a breast cancer patient. The study also has a pharmacoeconomic component.

DETAILED DESCRIPTION:
This study is a multi-center BCCA study that evaluates the impact of the Oncotype DX® assay on the decision making of the treating physician and the patient. The study also has a pharmacoeconomic component. All eligible patients in which either physician and/or patient determine that results from the 21 gene recurrence score could provide additional information useful in the decision making process regarding adjuvant chemotherapy or not will be asked by the participating physicians to participate in the study. If interested, the patient will consent to the study. The physician will complete a baseline questionnaire to document recommended adjuvant systemic therapies (pre-Oncotype DX®). The Oncotype DX® assay will be ordered after receipt of the Physician and Patient Registration and assignment of patient study number. The physician will discuss the results of the Oncotype DX® assay with the patient once the result is available and upon receipt of the pre-test questionnaire. The physician will complete a follow-up questionnaire (to document recommended adjuvant systemic therapies post Oncotype DX®) after the result of the Oncotype DX® assay is known.

ELIGIBILITY:
Inclusion Criteria:

1. Operable breast cancer with the primary tumour (pT1-3)
2. Pathological involvement (microscopic) of 1-3 lymph nodes. No minimum number of total lymph nodes need be resected. Extra-nodal extension of nodal deposit is allowed.
3. Her2Neu negative by IHC (0 or 1+) or FISH by current ASCO/CAP guidelines
4. Patient's tumor must undergo central review at GHI and there must be adequate material for the Oncotype DX® assay.
5. Patient's tumor must contain estrogen receptors (ER+).
6. Patient must be between the ages (inclusive) of 18-79.
7. Patient must be able to give informed consent
8. Patient has adequate performance status (PS ECOG 0,1 or Karnofsky ≥70) and be a medically fit candidate for treatment of their cancer with systemic chemotherapy in addition to hormonal therapy with no contra-indications to either systemic therapy maneuvers

Exclusion Criteria:

1. Patients have ER negative tumors (ER-) by local or central BCCA assessment
2. Patients have HER2 positive tumors by local or central BCCA assessment
3. Patients have four or more lymph node positive disease.
4. Lymph node involvement by isolated tumor cells or cells by IHC only (less than 200 cells and/or ≤0.2 mm)
5. Patients have known metastatic breast cancer.
6. Patients are unable to give consent or understand written language.
7. Patients with poor performance status (ECOG 2-4) in whom consideration of adjuvant chemotherapy or adjuvant hormonal therapy would be contraindicated.
8. Pregnant women in whom consideration of adjuvant chemotherapy or adjuvant hormonal therapy would be contraindicated.
9. Patients with tumors that on GHI central pathological review appears inadequate for the Oncotype DX® assay.

Ages: 18 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * 18-79 years old
  * Operative Primary Breast Cancer
    * Node + (N1-3: micrometastasis)
    * ER + and HER 2-
  * Candidate for adjuvant chemotherapy in addition to hormonal therapy
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-05; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Oncotype DX® assay affect on physician's treatment recommendations assessed by questionnaire | 1 Month
  The Oncotype DX® assay affect on physician's treatment recommendations pre and post Oncotype DX® Recurrence Score® result.

SECONDARY OUTCOMES:
Assessing Costs differences to the Publicly funded Health Care System | Data will be analyzed within 8 weeks of enrollment completion and presented within 9 months of study completion
  Costs to a publicly funded health care system

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Davidson JA, Cromwell I, Ellard SL, Lohrisch C, Gelmon KA, Shenkier T, Villa D, Lim H, Sun S, Taylor S, Taylor M, Czerkawski B, Hayes M, Ionescu DN, Yoshizawa C, Chao C, Peacock S, Chia SK. A prospective clinical utility and pharmacoeconomic study of the impact of the 21-gene Recurrence Score(R) assay in oestrogen receptor positive node negative breast cancer. Eur J Cancer. 2013 Jul;49(11):2469-75. doi: 10.1016/j.ejca.2013.03.009. Epub 2013 Apr 20. PMID 23611660